CLINICAL TRIAL: NCT05605119
Title: A Phase 1, Open Label, Dose Escalation, Dose Expansion, Multicenter, First in Human (FIH) Study Evaluating the Safety, Pharmacokinetics and Pharmacodynamics of Oral AUR105 in Patients With Relapsed Advanced Malignancies (SURYA-1)
Brief Title: First in Human, Dose Escalation, Dose Expansion Study of AUR105
Acronym: SURYA-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aurigene Discovery Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AUR105-101; CTRI/2022/09/046061 (Other: Clinical Trial registry of India)
Record Dates: First submitted 2022-10-05; First posted 2022-11-04 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor, Adult; Non-hodgkin Lymphoma; Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Intervention Model Description: Dose Escalation "3+3" dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AUR105 50mg to 750mg (Experimental): Currently planned dose levels in Part 1 are 50mg, 100mg, 200mg, 300mg, 450mg, 600mg and 740mg once daily
  Interventions: Drug: AUR105

INTERVENTIONS:
Drug: AUR105 — Once daily

SUMMARY:
This is a multi-center, open-label, First in Human, Phase 1 study of AUR 105 in adult patients with advanced malignancies.

The study will have two parts: a Dose Escalation Part and Dose Expansion Part.

DETAILED DESCRIPTION:
This is a Phase I, Open label First in Human Study in adult patients with relapsed advanced malignancies.

The study will have two parts. Dose escalation part and Dose expansion part

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1
* Acceptable bone marrow and organ function at screening as described below:

ANC ≥ 1500/μL (without WBC growth factor support) Platelet count ≥ 100,000/μL without transfusion support (Patients with lymphoma are allowed with Platelet count ≥ 75,000 / μL) Hemoglobin ≥ 9 g/dL (Transfusion is allowed to achieve this Hb) Total Bilirubin ≤ 1.5 x ULN; (Patients with known Gilbert's syndrome are allowed with a Total Bilirubin ≤ 2.5 x ULN) AST (SGOT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases) ALT (SGPT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases) Creatinine clearance (CrCl) ≥ 60 mL/min (either measured or estimated by the Cockcroft-Gault formula). (Cockcroft-Gault formula for estimated creatinine clearance [eCrCl]: eCrCl = [140- Age] × Weight [kg] × [0.85 if Female] / [72 × serum creatinine (mg/dL)]).

* Ability to swallow and retain oral medications
* Histo-pathological diagnosis of a solid tumor, Non-Hodgkin lymphoma or Hodgkin Lymphoma
* Evidence of measurable disease per RECIST, v1.1 for solid tumors (Eisenhauer et al. 2009) and per Lugano Criteria for Lymphoma (Cheson et al. 2014).
* Standard curative measures do not exist, and patient must have exhausted all effective therapies, available locally.

  1. At a minimum, solid tumor patients must have received at least two lines of systemic therapies in the metastatic incurable settings(these two lines must be in the metastatic setting and not in the earlier stage of cancer).
  2. At a minimum, lymphoma patients must have received at least 2 prior lines of systemic therapies. These systemic therapies could be either in the stage II, III or IV.

Exclusion Criteria:

* Systemic anti-cancer therapy, such as chemotherapy, or biological therapy, immunomodulatory drug therapy, received within the past 28 days or 5 half-lives, whichever is longer, from the Cycle 1 Day 1 of the study.
* Presence of an acute or chronic toxicity resulting from prior anticancer treatment, with the exception of alopecia or nail changes, that has not resolved to Grade ≤ 1, as determined by NCI CTCAE v 5.0
* Definitive Radiotherapy within the last 21 days of Cycle 1 Day 1 (limited field palliative radiation is allowed and no restrictions during the screening period or during the trial)
* Use of any investigational agent within 28 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1
* Use of moderate / strong CYP3A4 inhibitors/inducers or moderate / strong P-gp inhibitor/inducers within 2 weeks or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1 (The list of these medications is provided in the first four rows of Table 5)
* Known symptomatic or untreated or recently treated (≤ 6 months of screening) central nervous system (CNS) metastases or CNS lymphoma. Patients with previously treated (> 6 months of screening) CNS metastases or CNS lymphoma and are now stable and asymptomatic, from CNS perspective, are allowed
* Major surgery ≤ 28 days from Cycle 1 Day 1 (major surgery is defined as a procedure requiring general anesthesia)
* Patients with leukemia or myelodysplastic syndrome or multiple myeloma
* Active infection requiring systemic therapy.
* 10. Prophylactic use of antibiotics is allowed.
* Any infection detected during screening period which is resolved adequately according to investigator before the Cycle 1 Day 1, is allowed.
* Known to be human immunodeficiency virus (HIV) positive or have an acquired immunodeficiency syndrome-related illnessKnown active or chronic hepatitis B (HBsAg +ve) or hepatitis C infection (HCV antibody +ve)
* The patient who is expected to require any other form of antineoplastic therapy or targeted therapy while on study.
* Uncontrolled congestive heart failure (New York Heart Association [NYHA] Class 2-4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, or transient ischemic attack, or pulmonary embolism within 3 months prior to Cycle 1 Day 1
* Ongoing cardiac dysrhythmias requiring treatment of any grade or treatment of cardiac dysrhythmias in past 3 months, before Cycle 1 Day 1
* QTc (Bazzett) interval >450 ms for male patients or >460 ms for female patients on ECG at screening and/or at Cycle 1 Day 1 predose.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or significant gastritis, active bleeding diatheses, presence
* Current swab-positive or suspected (under investigation) Covid19 infection or fever and other signs or symptoms suggestive of Covid-19 infection with recent contact of person(s) with confirmed Covid-19 infection, at screening or Day 1 of Cycle 1
* History of another primary malignancy within 5 years prior to starting study drug, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study.
* Positive pregnancy test for women of child-bearing potential (WOCBP) at the screening or enrolment visit
* Lactating women or WOCBP who are neither surgically sterilized nor willing to use reliable contraceptive methods (hormonal contraceptive, IUD, or any double combination of male or female condom, spermicidal gel, diaphragm, sponge, cervical cap)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoints | 28 Days
  First cycle DLT
Primary Endpoints | Day 16
  PK parameters - Cmax
Primary Endpoints | Day 16
  PK parameters- AUC
Primary Endpoints | Day 16
  PK parameters- Tmax
Primary Endpoints | Through study completion, an average of 1 year
  Recommended Phase 2 Dose determination

SECONDARY OUTCOMES:
Exploratory Endpoints: | Day 15
  PD biomarkers (SDMA)
Exploratory Endpoints: | Through study completion, an average of 1 year
  Efficacy assessments overall response rate
Exploratory Endpoints: | Through study completion, an average of 1 year
  Efficacy assessments- duration of response
Exploratory Endpoints: | Through study completion, an average of 1 year
  Efficacy assessments- PFS
Exploratory Endpoints: | Through study completion, an average of 1 year
  Change in Tumor Specific Markers - CA-125 in ovarian cancer
Exploratory Endpoints: | Through study completion, an average of 1 year
  Change in Tumor Specific Markers - PSA in Castrate Resistant Prostate Cancer
Exploratory Endpoints: | Through study completion, an average of 1 year
  Change in Tumor Specific Markers - CEA in colorectal cancer

CONTACTS AND LOCATIONS:
Locations (9):
- India (9):
  - HCG City Cancer Center, Vijayawada, Andhra Pradesh
  - Omega Hospitals, Visakhapatnam, Andhra Pradesh
  - Kailash Cancer Hospital and Research Centre, Vadodara, Gujarat
  - Krupamayi Hospital, Aurangabad, Maharashtra
  - Moraya Multi-Speciality Hospital, Pune, Maharasthra
  - Sparsh Hospital and Critical Care, Bhubaneswar, Odisha
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - IMS&SUM Hospital, Bhubaneswar
  - ALL India Institute of medical Scieneces, New Delhi

IPD SHARING:
Plan to Share IPD: No